CLINICAL TRIAL: NCT06614608
Title: A Multi-Center, Randomized, Double-blind Phase I Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Efficacy of ASKC200 in Patients with Osteoarthritic Knee Pain
Brief Title: The Safety and Pharmacokinetics of ASKC200 in Osteoarthritic Knee Pain
Acronym: ASKC200
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu Aosaikang Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ASKC200-LC-102
Record Dates: First submitted 2024-09-13; First posted 2024-09-26 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Osteoarthritis, Knee; Pain
MeSH Terms: conditions — Osteoarthritis, Knee; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 5% ASKC200 (Experimental): A single dose will be topically applied to study knees for 60 minutes on Visit 1 on Day 1, Day 2, Day 3, and Day 4.
  Interventions: Drug: 5% ASKC200
- 1% ASKC200 (Experimental): A single dose will be topically applied to study knees for 60 minutes on Visit 1 on Day 1, Day 2, Day 3, and Day 4.
  Interventions: Drug: 1% ASKC200

INTERVENTIONS:
Drug: 5% ASKC200 — 5% ASKC200 is a multi-component formulation in which the active ingredient for the intended therapeutic effect is capsaicin at a level of 5% for this study.
  Arms: 5% ASKC200
Drug: 1% ASKC200 — 1% ASKC200 is a multi-component formulation in which the active ingredient for the intended therapeutic effect is capsaicin at a level of1% for this study.
  Arms: 1% ASKC200

SUMMARY:
This is a multi-center, randomized, double-blind clinical trial to evaluate the safety, tolerability, pharmacokinetics, and efficacy of ASKC200 in subjects with OA of the knees and determine the phase II recommended dose. Assigned doses will be applied for 60 minutes on each of four consecutive days.

DETAILED DESCRIPTION:
Subjects will be randomized to one of the two Arms in this study: 5% ASKC200 or 1% ASKC200. All subjects will receive 4 consecutive days of treatment and will then be followed up until the Day 34 visit.

The NRS score of weekly average of average daily pain intensity (WAADPI) of the study knee should ≥ 5 and the NRS score of WAADPI of the contralateral knee should < 4 at screening.

Data will be collected from Day 1 through Day 5 and then again on Days 19 and 34 for efficacy, tolerability, and safety measures.

ELIGIBILITY:
Inclusion Criteria:

1. Sign informed consent prior to any inspection and evaluation, and understand and follow test requirements;
2. Age 40-75 years old (including boundary value) at the time of signing the informed consent, gender is not limited;
3. Primary knee osteoarthritis was confirmed by clinical and imaging examination;
4. Knee osteoarthritis pain history ≥6 months;
5. Tibial joint X-ray within 3 months prior to drug administration showed that the tibiofemoral joint of the target knee was graded Kellgren-Lawrence II or III;
6. Before the first medication, the WAADPI NRS score of the study knee was ≥5, and the WAADPI NRS score of the contralateral knee was <4;
7. Be willing to discontinue the use of nonsteroidal anti-inflammatory drugs, acetaminophen, and other pain medications, and only use the acetaminophen provided in the study for emergency treatment of knee osteoarthritis pain during the study period;
8. Body mass index (BMI) ≤40.0 kg/m2.

Exclusion Criteria:

1. Secondary arthritis caused by other causes;
2. The study knee has other knee pathologic findings confirmed by clinical evaluation or imaging
3. There are other conditions that can cause study knee pain or other physical pain;
4. Other medications for osteoarthritis were used within 1 week prior to the first dose;
5. Patients with chronic pain in other parts of the body requiring long-term oral analgesic therapy, or those requiring combined treatment with systemic glucocorticoids;
6. Open knee injury or knee surgery occurred in the study knee within 6 months before the first medication; Or have had any major surgical procedures within 3 months prior to the first medication;
7. The study knee has received intra-articular injection treatment (such as steroids or sodium hyaluronate, etc.) within 3 months before the first medication;
8. Received physical therapy for study knee osteoarthritis (such as electrotherapy or acupuncture) within 3 months before the first medication;
9. Used any capsaicin-containing product or non-steroidal anti-inflammatory drug on the knee within 2 weeks prior to the first administration;
10. Have An open wound, skin erythema or edema, skin infection, or any other skin lesion in the study knee prior to initial administration;
11. A history of alcohol or drug dependence within 12 months prior to the first administration or a positive urine drug test during the screening period.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Safety:Incidence of adverse events（AEs） | 34 days
  All adverse medical events occurring after the subject receives the investigational drug, which may be manifested as symptoms, signs, diseases, or abnormalities in laboratory tests, but may not necessarily have a causal relationship with the investigational drug.

SECONDARY OUTCOMES:
Efficacy:Change in the NRS score of weekly average of average daily pain intensity(WAADPI) From Baseline | Day 19, Day 34
  The average amount of pain as reported by the subject using a 0 - 10 numerical rating scale (NRS). Higher scores indicate more pain.
Efficacy:Remission ratio of study knee according to NRS score | Day 19, Day 34
  The average amount of pain as reported by the subject using a 0 - 10 numerical rating scale (NRS). Higher scores indicate more pain.
Efficacy:Change in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Score From Baseline | Day 19, Day 34
  The WOMAC Index is a questionnaire used to assess health status and health outcomes in KOA. The questionnaire contains 24 questions（0-10） on pain, stiffness and physiology, will ask participants to complete the WOMAC questionnaire considering their symptoms in the past 48 hours.Higher scores indicate more pain.
Efficacy:Change in patients clinical general impression (PCGI-C) | Day 19, Day 34
  The change in patients clinical general impression as reported by the subject using a 0 - 7 scale (PCGI-C).Higher scores indicate worse state of pain.
Efficacy:The use of acetaminophen | 34 days
  Subjects will record their administration of acetaminophen . The number of days the subjects use acetaminophen and the proportion of subjects who use acetaminophen will be counted.
Maximum Observed Plasma Concentration (Cmax) for ASKC200 | Day1-Day5
Time of First Occurrence of Cmax (Tmax) for ASKC200 | Day1-Day5
Area Under the Plasma Concentration-time Curve from Time 0 to 24 Hours (AUC24) for for ASKC200 | Day1-Day5

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Hospital, Beijing, Beijing Municipality, China